CLINICAL TRIAL: NCT04580693
Title: The Impact of Exercise-Induced Cardiac Remodeling on Myocardial Efficiency: A Multimodality Structural, Functional, and Metabolic Evaluation.
Brief Title: The Impact of Exercise-Induced Cardiac Remodeling on Myocardial Efficiency
Status: Completed | Type: Observational
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Brigham and Women's Hospital (Other); National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Meagan Murphy Wasfy, Principal Investigator, Massachusetts General Hospital
Other Study IDs: 2014P000781; K23HL136902 (NIH)
Record Dates: First submitted 2020-09-28; First posted 2020-10-08 (Actual); Last update posted 2025-05-16 (Actual); Status verified 2025-05

CONDITIONS: Cardiomyopathy, Hypertrophic
Keywords: Cardiomyopathy, Hypertrophic; Athletes, Endurance; Healthy Volunteers
MeSH Terms: conditions — Cardiomyopathy, Hypertrophic | interventions — Magnetic Resonance Spectroscopy

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Blood draws for analysis of blood for metabolic parameters (glucose, insulin, and free fatty-acid levels).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- Healthy Volunteers/Control: Age and body surface area (BSA) matched volunteers who are sedentary or normally active. Normally active is defined as less than 5 hours of exercise per week. Healthy volunteer subjects must be able to exercise on an upright bicycle ergometer and be between the ages of 18-50.
  Interventions: Other: PET Scan
- Hypertrophic Cardiomyopathy/HCM: HCM subjects are patients that are age and BSA-matched with the athletes who then have an established clinical diagnosis of HCM without left ventricular (LV) outflow tract obstruction. There can be no anticipated changes to baseline exercise program (if any) over the study period. HCM subjects must be able to exercise on an upright bicycle ergometer and be between the ages of 18-50.
  Interventions: Other: PET Scan
- Endurance Athletes: Official participation in a collegiate athletic varsity rowing team OR participation in competitive endurance athletics. Competitive endurance athletics is defined as greater than or equal to 10 hours of exercise training per week with the majority dedicated to endurance activities such as cycling, rowing, or running. Endurance athlete subjects must be able to exercise on an upright bicycle ergometer and be between the ages of 18-50.
  Interventions: Other: PET Scan

INTERVENTIONS:
Other: PET Scan — PET scan using a tracer that is under a physician sponsored IND.

SUMMARY:
This research study is being conducted to find out how heart function and energy use differ among healthy endurance athletes, individuals who do not exercise regularly, and patients with hypertrophic cardiomyopathy. The research study involves taking part in a cardiopulmonary exercise test (CPET), two positron emission tomography (PET) scans, an echocardiogram, and blood draws. The study will consist of a total of three visits scheduled over a maximum of two weeks. By determining how heart function and energy use differ between our three groups of healthy endurance athletes, individuals who do not exercise regularly, and patients with hypertrophic cardiomyopathy, the investigators hope to have this work translate into a novel clinical tool for differentiating pathologic changes of the heart from physiological changes in heart. This is otherwise known as "gray-zone" left ventricular hypertrophy, or enlargement of the left ventricle.

DETAILED DESCRIPTION:
The investigators anticipate that by defining the myocardial metabolic profiles of exercise-induced left ventricular hypertrophy (EI-LVH) and hypertrophic cardiomyopathy (HCM), we will determine if these differ sufficiently to distinguish these two forms of LVH. Because HCM causes sudden death with physical activity, it is critically important to determine the etiology of undifferentiated "gray zone" LVH in the athlete presenting for medical evaluation, and existing mechanisms of assessing myocardial structure and function are not universally adequate. The investigators anticipate that the work may translate into a novel clinical tool for differentiating pathology from physiology in "gray-zone" LVH. The complementary mechanistic goal of this study is to combine comprehensive evaluations of myocardial functional parameters and metabolism to better understand the link between function and metabolism and, ultimately, the biological mechanisms of EI-LVH and LVH due to HCM. There are three specific aims to the research study. The first specific aim is to define the relationships between changes in myocardial metabolic efficiency (MME) and changes in myocardial mechanics that accompany EI-LVH. The second is to establish and compare myocardial metabolic profiles of EI-LVH and HCM. The third is to analyze a subset of the endurance athlete subjects to determine the impact of aerobic exercise training on MME over a 90-day period.

The study will employ a mixed study design. The study is a cross-sectional design but will analyze a subset of endurance athletes longitudinally with repeated measures after 90 days from the first three study visits.

For the cross sectional design, the first study visit will be at Massachusetts General Hospital and will involve a cardiopulmonary exercise test (CPET) on an upright bicycle, with blood sampling before the CPET at rest, and after exercise. Study visits two and three will follow the same protocol. Both study visits two and three will occur at Brigham and Women's Hospital and will involve an echocardiogram and a positron emission tomography (PET) scan. Both visits will include blood sampling at rest, and then either the resting PET scan or a PET scan after acute exercise provocation on a supine bicycle. Study visits two and three will occur on two sequential mornings.

ELIGIBILITY:
Inclusion Criteria for Endurance Athletes:

* Age ≥ 18-60
* Official participation in a collegiate varsity rowing team OR participation in competitive endurance athletics (defined as >= 10 hours of exercise training per week with the majority dedicated to endurance activities (i.e. cycling, rowing, running).

Inclusion Criteria for Healthy Volunteers:

* Age ≥ 18-60
* 0-5 hours of exercise per week without anticipated changes in exercise habits over study period
* Able to exercise on an upright bicycle ergometer

Exclusion Criteria for Endurance Athletes and Healthy Volunteers:

* Known medical disease (including but not limited to known cardiac or pulmonary disease, diabetes or contraindications to exercise testing such as uncontrolled cardiac arrhythmia, excessive blood pressure of more than 200/100 mmHg at rest, active exacerbation of congestive heart failure or reactive airways disease).
* Pregnancy

Inclusion Criteria for HCM Patients:

* Established HCM diagnosis as per above (20 subjects)
* Age ≥ 18-50
* No anticipated changes to baseline exercise program (if any) over the study period
* Able to exercise on an upright bicycle ergometer

Exclusion Criteria for HCM Patients:

* Obstructive LVOT gradient > 30 mmHg, at rest or with provocation.
* Reduced LVEF < 53%.
* NYHA class III or IV heart failure symptoms.
* History of sudden cardiac death or hemodynamically significant ventricular tachycardia.
* History of unexplained syncope.
* Having a Class I or IIa AHA/ACC indication for ICD placement without an ICD
* Known medical disease (including but not limited to known cardiac or pulmonary disease other than HCM, diabetes, or contraindications to exercise testing such as uncontrolled cardiac arrhythmia, excessive blood pressure of more than 200/100 mmHg at rest, active exacerbation of congestive heart failure or reactive airways disease).
* Pregnancy

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Endurance Athletes: A collegiate rowing team or invitation to participate from local endurance type athletic clubs. (i.e. running clubs, rowing teams, etc.) HCM Patients: MGH Hypertrophic Cardiomyopathy Program's database, the Research Patient Data Registry (RPDR), and through the BWH Hypertrophic Cardiomyopathy Program's patient panel. Also RALLY.
  Healthy Control/Volunteers: Partners RALLY (research ally) website.
Sampling Method: Non-Probability Sample
Enrollment: 87 (Actual)
Dates: Start 2019-02-28 (Actual); Primary Completion 2022-06-09 (Actual); Study Completion 2022-06-09 (Actual)

PRIMARY OUTCOMES:
Myocardial Metabolic Efficiency | up to 2 weeks
  The ratio of myocardial oxygen consumption to myocardial work.

SECONDARY OUTCOMES:
Myocardial Blood Flow Reserve using PET | up to 2 weeks
  Difference in blood flow at rest and with exercise.

OTHER OUTCOMES:
Left Ventricular Mass | up to 2 weeks
  Size of the left ventricle.

CONTACTS AND LOCATIONS:
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No